CLINICAL TRIAL: NCT06481319
Title: Implementing a Pilot Patient Navigator Program to Improve Access to Infertility Care for Underserved Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-44747
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Infertility
Keywords: Infertility Patient Navigator (PN); Under-resourced patients; Cycle based testing; Urology appointments; Health Literacy; Boston Medical Center
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: One group intervention with age-matched historical controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infertility Patient Navigator Group (Experimental): Participants in this group will receive assistance from the Infertility Patient Navigator (PN) to schedule and complete the infertility evaluation.
  Interventions: Behavioral: Infertility Patient Navigator
- Historical Comparison Group (No Intervention): Age-matched controls selected from the electronic medical record database who received infertility evaluation without PN assistance.

INTERVENTIONS:
Behavioral: Infertility Patient Navigator — Assistance with infertility evaluation including scheduling appointments
  Arms: Infertility Patient Navigator Group

SUMMARY:
This investigators will conduct a pilot study investigating the implementation of an infertility Patient Navigator (PN) program to mitigate challenges for underserved individuals at Boston Medical Center (BMC) seeking infertility care. The primary objective is to assess whether the PN program can significantly reduce time to completion of infertility evaluation and to initiation of fertility treatment (if recommended) for infertile patients from an underserved patient population.

The study aims are to:

1. evaluate the impact of the PN program on timelines including obtaining commercial insurance coverage for infertility, expediting labwork/imaging, weight management, and partner urology appointments, and initiating fertility treatment; and
2. ascertain the medical literacy of participants with a validated tool to assess the impact of low medical literacy on PN facilitation.

Participants will be contacted by the PN and provided with a survey instrument that will test their medical literacy. Then the PN will assist with scheduling cycle-based testing including labwork and uterine cavity evaluation, the partner's urology appointment, the patient's appointments such weight management/nutrition referral, mammograms (if indicated by age), and insurance counseling if the participant's current insurance does not cover infertility diagnostic testing and treatment. These tasks are part of pursuing fertility care at BMC.

Duration of evaluation and time to treatment in age-matched control patients from the year prior that did not have PN services will be utilized as a comparison group.

Regression analyses will be conducted to explore the association between utilization of a PN and pregnancy rates, considering potential confounding factors.

Establishment of the pilot program will enable the investigators to apply for a larger institutional patient care grant going forward. Strategies developed through this research can may enhance fertility care access for underserved communities across various healthcare settings. By tailoring interventions to populations not usually able to access specialized healthcare services, this study pioneers a paradigm shift towards inclusivity and equity in reproductive medicine.

ELIGIBILITY:
Inclusion Criteria:

Intervention cases

* A new patient at BMC Reproductive Endocrinology for the diagnosis of infertility from July 1, 2024 to January 31, 2025 Controls
* A new patient at BMC Reproductive Endocrinology for the diagnosis of infertility from July 1, 2023 to January 31, 2024.

Exclusion Criteria:

* Patients in whom fertility treatment with their own eggs is not recommended, egg freezing or oncofertility cycles.
* Non-English speaking

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Time to complete infertility evaluation | 12 months
  This outcome will be assessed by data abstracted from the electronic medical record (EMR).
Time to start fertility treatments | 12 months
  This outcome will be assessed by data abstracted from the EMR.
Wait time for urology appointments | 12 months
  This outcome will be assessed by data abstracted from the EMR.
Wait time for weight management appointments | 12 months
  This outcome will be assessed by data abstracted from the electronic medical record.

SECONDARY OUTCOMES:
Pregnancy rate | 12 months
  This outcome will be assessed by data abstracted from the EMR by dividing the number of pregnancies by the number of participants.
Time to live birth | 12 months
  This outcome will be assessed by data abstracted from the EMR.
Frequency of PN contacts in Intervention Group | 12 months
  This outcome will be assessed from data documented by the PN study records for each participant in the Intervention group
Number of PN contacts in Intervention Group | 12 months
  This outcome will be assessed from data documented by the PN study records for each participant in the Intervention group
Duration of PN contacts in Intervention Group | 12 months
  This outcome will be assessed from data documented by the PN study records for each participant in the Intervention group

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Kuohung, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Reproductive Endocrinology, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No